CLINICAL TRIAL: NCT02972723
Title: A Study of the Antiviral Activity of Metformin as an Anti-Hepatitis C Virus Agent in Patients With Chronic Hepatitis C Virus Infection
Brief Title: Metformin Therapy in HCV Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 10ID003; 2010-022850-18 (EudraCT Number)
Record Dates: First submitted 2016-10-27; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Metformin Therapy in HCV
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin therapy, single arm (Experimental): Open label trial, participants will be expected to take Metformin twice a day for 2 weeks
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Oral Metformin 1g bd. (total = 2g per day) for 14 days
  Other Names: Glucophage

SUMMARY:
Hepatitis C virus infection (HCV) is a major cause of cirrhosis and death from liver disease worldwide. Current therapy for HCV with interferon based therapies results in cure rates of around 5055% which leaves a significant number of patients without effective therapy. HCV induces (can bring on) insulin resistance and insulin resistance is a factor known to reduce the response to antiHCV therapy. This finding stimulated initial studies looking at agents that may reduce insulin resistance as additional therapy in HCV infection.

A study using metformin in addition to interferon and ribavirin showed a nonsignificant increase in cure rates (53% vs. 42%), but this was limited to patients with type 1 infection AND demonstrable insulin resistance. The assumption was made that the potential effect of metformin was likely to be on insulin resistance and thus by modulating this enhances response. The investigators (Prof M Harris, University of Leeds) have data (currently unpublished)suggesting that metformin may have an antiviral effect independent of its effect on insulin resistance, thus raising the possibility that metformin may have a direct antiviral effect in vivo. Given that the development of specific antiHCV agents which target viral proteins such as its polymerase and protease are in trial development but have so far proved either highly toxic or are likely to have a huge cost there is considerable rationale for looking at alternative potential antiHCV agents and in this context metformin is cheap, readily available and has an excellent safety profile. This pilot study therefore addresses the question "Does metformin therapy result in a significant drop in HCV viral load in chronically infected patients?"

ELIGIBILITY:
Inclusion Criteria:

* Adult Males and Females (18-70 yrs old) able to give consent
* Chronic hepatitis C virus infection
* Women of child bearing potential (who have a negative pregnancy test) must agree to use methods of medically acceptable forms of contraception during the study; (e.g.intra-uterine device (IUD) or a double-barrier method of oral contraception with condom)

Exclusion Criteria:

* Type 2 diabetes.
* Patients with impaired renal function.
* Decompensated liver cirrhosis (stable patients with cirrhosis would be eligible).
* Patients who in the opinion of the Investigator are considered unsuitable.
* Pregnant females.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Drop of viral load by at least 1 log in patients receiving Metformin | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Dr Ryder, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Secondary care Hepatitis clinic at Nottingham University Hospital, Nottingham, Nottingham, United Kingdom